CLINICAL TRIAL: NCT04495829
Title: Clinical and Refractive Outcomes After Contoura® Refractive Surgery Planned Using Phorcides Surgery Planning Software
Status: Completed | Type: Observational
Sponsor: American Corneal Consultants (Other)
Collaborators: Science in Vision (Other); Alcon Research (Industry)
Responsible Party: Sponsor
Other Study IDs: ML-2020-01
Record Dates: First submitted 2020-07-27; First posted 2020-08-03 (Actual); Results first posted 2022-04-14 (Actual); Last update posted 2023-07-20 (Actual); Status verified 2022-02

CONDITIONS: Refractive Errors
MeSH Terms: conditions — Refractive Errors

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Phorcides: Both eyes of subjects eligible for Contoura(R) topography-guided ablation with the Wavelight excimer laser, with surgery planned using Phorcides software.
  Interventions: Device: Phorcides Analytical Engine

INTERVENTIONS:
Device: Phorcides Analytical Engine — Surgery planning using the Phorcides analytical engine.
  Other Names: Phorcides

SUMMARY:
The objective of the current study is to prospectively evaluate 3-month clinical outcomes from LASIK performed using the Phorcides surgical planning software with Contoura topography-guided ablation in both eyes of subjects with myopia and myopic astigmatism seeking refractive surgery for distance correction.

DETAILED DESCRIPTION:
The objective of the current study is to prospectively evaluate 3-month clinical outcomes from LASIK performed using the Phorcides surgical planning software with Contoura topography-guided ablation in both eyes of subjects with myopia and myopic astigmatism seeking refractive surgery for distance correction. Data will be compared to published results for wavefront optimized LASIK and LASIK performed with Contoura using other refractive algorithms.

The hypothesis is that use of the Phorcides planning software will result in a higher percentage of eyes with residual refractive cylinder ≤ 0.25D than will be achieved with wavefront-optimized (WFO) LASIK. It is also expected that unaided postoperative visual acuity and visual symptoms will be improved.

ELIGIBILITY:
Inclusion Criteria:

* Candidate for Contoura excimer laser vision correction
* Gender: males and females.
* Age: 20 or older
* Willing and able to provide written informed consent for participation in the study.
* Willing and able to comply with scheduled visits and other study procedures.
* Good ocular health, with no pathology that compromises visual acuity (other than refractive error)
* Corrected preoperative visual acuity of 20/20 (0.0 logMAR) or better in the eye being treated
* Meet Contoura eligibility requirements (approved range): up to -8.00 D sphere, up to -3.00 D cylinder, and a spherical equivalent no greater than -9.00 D
* Desire good vision at distance in both eyes

Exclusion Criteria:

* Corneal pathology (e.g. opacities, epithelial basement membrane dystrophy, Fuchs' dystrophy, etc.)
* Previous corneal surgery (e.g., radial keratotomy, corneal refractive surgery or corneal transplant, DSAEK, DMEK, lamellar keratoplasty)
* Previous anterior or posterior chamber surgery (e.g., vitrectomy, laser iridotomy)
* Desire for good uncorrected near vision in one or both eyes
* Participation in (or current participation) any investigational drug or device trial within the previous 30 days prior to the start date of this trial
* Unsuitability for the trial, in the opinion of the investigator, for any reason
* Pregnancy or desire to become pregnant during the trial
* Intraoperative complications.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy subjects presenting for myopic LASIK correction who are eligible for treatment with topography-guided ablation in both eyes.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2020-07-24 (Actual); Primary Completion 2021-04-21 (Actual); Study Completion 2021-04-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert D Stulting, Principal Investigator — Woolfson Eye Institute
Locations (5):
- United States (5):
  - Woolfson Eye Institute, Atlanta, Georgia
  - North Suburban Eye Specialists, Coon Rapids, Minnesota
  - TLC Laser Eye Center, Chesterfield, Missouri
  - Laser Defined Vision, Greensboro, North Carolina
  - Mann Eye Institute and Laser Centers, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Stulting RD, Durrie DS, Potvin RJ, Linn SH, Krueger RR, Lobanoff MC, Moshirfar M, Motwani MV, Lindquist TP, Stonecipher KG. Topography-Guided Refractive Astigmatism Outcomes: Predictions Comparing Three Different Programming Methods. Clin Ophthalmol. 2020 Apr 24;14:1091-1100. doi: 10.2147/OPTH.S244079. eCollection 2020. PMID 32425495
- [Result] Lobanoff M, Stonecipher K, Tooma T, Wexler S, Potvin R. Clinical outcomes after topography-guided LASIK: comparing results based on a new topography analysis algorithm with those based on manifest refraction. J Cataract Refract Surg. 2020 Jun;46(6):814-819. doi: 10.1097/j.jcrs.0000000000000176. PMID 32176160
- [Derived] Stulting RD, Lobanoff M, Mann PM 2nd, Wexler S, Stonecipher K, Potvin R. Clinical and refractive outcomes after topography-guided refractive surgery planned using Phorcides surgery planning software. J Cataract Refract Surg. 2022 Sep 1;48(9):1010-1015. doi: 10.1097/j.jcrs.0000000000000910. PMID 35171146

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Phorcides
Started | 70
Completed | 65
Not Completed | 5
Not completed — Lost to Follow-up | 2
Not completed — Inclusion criterion not met | 3

BASELINE CHARACTERISTICS:
Units Other Than Participants: Eyes
Arm/Group | Phorcides
Number analyzed (Participants) | 70
Number analyzed (Eyes) | 140
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Only subjects competing the 3-month visit were included
  years
    number analyzed (Participants) | 65
    (all) | 31 (5.4)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Only subjects completing the 3-month visit are included
  Participants
    number analyzed (Participants) | 65
    Female | 38
    Male | 27
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
  Participants
    number analyzed (Participants) | 0
Region of Enrollment [Number; unit: participants]
  United States | 70
MRSE [Mean (Standard Deviation); unit: diopters] | -3.6 (1.79)
Refractive cylinder [Mean (Standard Deviation); unit: diopters] | 0.54 (.49)
Uncorrected distance VA [Mean (Standard Deviation); unit: logMAR (log of min angle of resolution] | .95 (.33)
Corrected distance VA [Mean (Standard Deviation); unit: logMAR] | -.04 (.04)

OUTCOME MEASURES:

1. Primary Outcome: Residual Refractive Cylinder
Description: Residual refractive cylinder in diopters
Time Frame: 3 months postop
Measure: Mean (Standard Deviation); unit: diopters
Units Other Than Participants: Eyes
Arm/Group | Phorcides
Number analyzed (Participants) | 65
Number analyzed (Eyes) | 130
diopters | 0.04 (0.09)

2. Secondary Outcome: Uncorrected Distance Visual Acuity
Description: Uncorrected visual acuity at distance (4-6m)
Time Frame: 3 months postop
Measure: Mean (Standard Deviation); unit: logMAR
Units Other Than Participants: Eyes
Arm/Group | Phorcides
Number analyzed (Participants) | 65
Number analyzed (Eyes) | 130
logMAR | -.11 (0.06)

3. Secondary Outcome: Residual Refractive Sphere
Description: Residual refractive spherical equivalent in diopters
Time Frame: 3 months postop
Measure: Mean (Standard Deviation); unit: diopters
Units Other Than Participants: Eyes
Arm/Group | Phorcides
Number analyzed (Participants) | 65
Number analyzed (Eyes) | 130
diopters | 0.08 (0.20)

4. Secondary Outcome: Satisfaction and Vision
Description: A questionnaire related to visual quality and satisfaction after surgery
Time Frame: 3 months postop
Measure: Count of Participants; unit: Participants
Arm/Group | Phorcides
Number analyzed (Participants) | 65
Participants
  Double vision: None to moderate | 65
  Double vision: Marked to severe | 0
  Trouble driving at night: None to moderate | 65
  Trouble driving at night: Marked to severe | 0
  Trouble reading: None to moderate | 65
  Trouble reading: Marked to severe | 0
  Dryness: None to moderate | 63
  Dryness: Marked to severe | 2
  Foreign body sensation: None to moderate | 65
  Foreign body sensation: Marked to severe | 0
  Fluctuation in vision: None to moderate | 65
  Fluctuation in vision: Marked to severe | 0
  Glare: None to moderate | 65
  Glare: Marked to severe | 0
  Halos: None to moderate | 65
  Halos: Marked to severe | 0
  Light sensitivity: None to moderate | 63
  Light sensitivity: Marked to severe | 2
  Pain: None to moderate | 65
  Pain: Marked to severe | 0
  Starbursts: None to moderate | 65
  Starbursts: Marked to severe | 0

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Phorcides
All-Cause Mortality (participants affected / at risk) | 0/70
Serious Adverse Events (participants affected / at risk) | 0/70
Other Adverse Events (participants affected / at risk) | 1/70
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phorcides (N=70)
Epithelial defect (Eye disorders) | 1 (1) — Epithelial defect

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-07-15): https://cdn.clinicaltrials.gov/large-docs/29/NCT04495829/Prot_SAP_000.pdf